CLINICAL TRIAL: NCT03087136
Title: A Multicenter Observational Study to Evaluate Pediatric Multiple Sclerosis in Brazil
Acronym: EMOCEMP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Other Study IDs: 61080516.4.1001.5336
Record Dates: First submitted 2017-03-15; First posted 2017-03-22 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; pediatric
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: anti-aquaporin-4 antibody — Serum anti-aquaporin-4 antibody
Diagnostic Test: anti-myelin oligodendrocyte glycoprotein — Serum anti-myelin oligodendrocyte glycoprotein
  Other Names: (anti-MOG)

SUMMARY:
Pediatric Multiple sclerosis (MS) is a chronic inflammatory disease defined by multiple episodes of demyelination of the central nervous system (CNS) separated by time and space as specified in adults not explained by acute disseminated encephalomyelitis (ADEM). Several studies have indicated that at least 5% of MS patients are in the pediatric population, but no prospective study was performed in Brazil. There are particular characteristics of Pediatric MS that differs from the adult population and have been focus of interest in the last years. However, we still lack high evidence data, specially concerning treatment, of this age group.

This is an observational non-interventional multicenter study in pediatric MS patients in which participating subjects will be characterized by their clinical, MRI and immunological features. In this observational study, we will select 8 MS centers in Brazil to recruit at least 100 pediatric patients currently followed on each center with idiopathic inflammatory CNS disorders over a 2-year study period. We will collect retrospective and prospective clinical and MRI data to determine the proportion of patients who fulfill the International Pediatric Multiple Sclerosis Study Group (IPMSSG) criteria for MS,7 especially on those below 10 years where the use of McDonald 2010 criteria is not recommended routinely. Following the inclusion on the study, subjects will be followed for at least 2 years.

All subjects enrolled in this study will have serum collected to test autoantibodies including anti-AQP4 and anti-MOG using cell-based assays with transfected cells.8 Pediatric patients with positive testing for these autoantibodies will be analyzed separately.

Exploratory MRI sub-study In 10 patients recruited at Hospital São Lucas PUCRS, we will perform an exploratory substudy with advanced MRI using q-space diffusion protocol on a 3-Tesla MRI (GE Signa HDx 3.0T, General Electric, Milwaukee, WI, USA) and a 8-channel head coil to visualize remyelinating brain MS lesions. Normalized leptokurtic diffusion (NLD) data will be acquired using diffusion-weighted echo planar imaging. All MRI scans from this exploratory study will be performed at the Brain Institute of Rio Grande do Sul (BraIns). Only patients with previous brain demyelinating lesions will be included in this exploratory sub-study.

ELIGIBILITY:
Inclusion Criteria:

1. Parents / patient have an understanding, ability and willingness to fully comply with study procedures
2. Parents / patient have the ability to provide voluntary written, signed and dated informed consent to participate in the study
3. Be 6 months - 18 years of age at screening
4. Have clinical evidence of at least 1 attack suggestive of idiopathic inflammatory CNS disorder
5. Have at least one brain MRI with available images (for review)

   * For the exploratory MRI study, parents / patients have to agree to perform 2 MRI scans (at baseline and at the end of the study). Considering the age of the study subjects, sedation may be required during the acquisition of the MRI.

Exclusion Criteria:

1. Current evidence or known history of clinically significant infection including:

   - Chronic or ongoing active infectious disease requiring long-term systemic treatment such as active hepatitis B or C, HIV or tuberculosis
2. Current malignancy or history of malignancy in the past 5 years
3. Significant concurrent, uncontrolled medical condition that could affect subject's safety or impair the subject's participation in the study.
4. Current participation in any interventional trial.
5. Pregnant or breastfeeding

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In this observational study, we will select 8 MS centers in Brazil to recruit at least 100 pediatric patients currently followed on each center with idiopathic inflammatory CNS disorders over a 2-year study period.
  We will collect retrospective and prospective clinical and MRI data to determine the proportion of patients who fulfill the International Pediatric Multiple Sclerosis Study Group (IPMSSG) criteria for MS, especially on those below 10 years where the use of McDonald 2010 criteria is not recommended routinely. Following the inclusion on the study, subjects will be followed for at least 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Convertion rate to MS | 2 years
  To evaluate the proportion of patients (below and above 10 years-old) with idiopathic inflammatory CNS disorders converting to pediatric MS in Brazilian MS referral centers.

SECONDARY OUTCOMES:
Clinical features | 2 years
  • To compare the clinical and MRI features between pediatric MS patients with disease onset < 10 and > 10 years
epidemiology | 2 years
  • To analyze the influence of latitude, ethnicity and past viral infections on the development of pediatric MS
autoantibodies | 2 years
  • To determine the proportion of patients with pediatric MS and other inflammatory demyelinating CNS disorders with autoantibodies (anti-AQP4 and anti-MOG)
treatments | 2 years
  • To identify the disease-modifying treatments used in pediatric MS cases by the treating physician and the occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Sato, Principal Investigator — Pontifical Catholic University of Rio Grande do Sul
Locations (8):
- Brazil (8):
  - Universidade Federal de Uberlândia, Uberlândia, Minas Gerais
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Hospital da Restauração de Recife, Recife, Pernambuco
  - Universidade Federal do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Pontifical Catholic University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto / Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No